CLINICAL TRIAL: NCT04925518
Title: Closed Loop Mechanical Ventilation Coupled to Extracorporeal Membrane Oxygenation Support in Therapy Refractory Acute Respiratory Distress Syndrome and Cardiogenic Shock
Brief Title: Closed Loop Mechanical Ventilation and ECMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ECMO - IV
Record Dates: First submitted 2021-05-31; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Acute Respiratory Distress Syndrome; Cardiogenic Shock
Keywords: ECMO; ECLS; Mechanical Ventilation; Lung Protective Ventilation; Closed Loop Ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock, Cardiogenic

STUDY DESIGN:
Intervention Model Description: Patients are initially mechanically ventilated with a conventional mechanical ventilation mode after ECMO installation, once steady state on the conventional mode is achieved for several hours, switch to the closed loop ventilation mode.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Ventilation Mode (Active Comparator): Patients mechanically ventilated with a conventional mechanical ventilation mode until steady state is achieved for several hours.
  Interventions: Device: Conventional Mechanical Ventilation
- Closed Loop Ventilation Mode (Experimental): Once steady state on the conventional mechanical ventilation mode is achieved for several hours, switch to closed loop ventilation mode for the remainder of the study period.
  Interventions: Device: Closed Loop Mechanical Ventilation

INTERVENTIONS:
Device: Closed Loop Mechanical Ventilation — Closed loop ventilation mode (Intellivent-ASV+®). Intellivent-ASV+® was initiated by activating the controllers for minute volume, PEEP (range 5 to 18 cmH2O) and fraction of inspired oxygen (FiO2) (range 21 to 100 %). The target shift ranges for CO2-management were set between -2.5 and +2.5 kPa, and for O2-management between -2 and +2 %.
  Other Names: Intellivent-ASV+®
  Arms: Closed Loop Ventilation Mode
Device: Conventional Mechanical Ventilation — Mechanical ventilation with a conventional mode, usually either biphasic positive airway pressure ventilation (DuoPAP®) or adaptive support ventilation (ASV®)
  Other Names: DuoPaP/ ASV
  Arms: Conventional Ventilation Mode

SUMMARY:
Mechanical ventilation and ECMO are both technologies interacting on gas exchange. Nevertheless, besides a consensus paper, no evidence-based guidelines regarding protective lung ventilation on ECMO exist to date. Mechanical Ventilation with Intellivent-ASV, an algorithm driven, closed loop system, provides an opportunity to standardize ventilation on ECMO.

We propose and validate lung protective ventilation with a closed loop ventilation mode in patients with ECMO.

DETAILED DESCRIPTION:
In critically ill patients admitted to the intensive care unit due to either acute respiratory failure or circulatory collapse, mechanical ventilation in combination with either extra-corporal lung assist (VV ECMO) or cardiac assist (VA ECMO) is increasingly used. Both mechanical ventilation and ECMO contribute to the control of gas exchange hence need to be adjusted accordingly.

As an assist device like a VV ECMO or a VA ECMO the control the gas exchange needs to be adjusted via sweep gas flow (ventilation), fraction of oxygen in the sweep gas (oxygenation, FsO2) and blood flow over the extracorporeal device. The combination of adaptive ventilation with ECMO is a novel concept allowing the control of oxygenation and ventilation by the adjustment of the ECMO device only.

Adaptive lung ventilation is a category of ventilation modes, which allow the control of oxygenation and ventilation with a closed loop. Using this type of ventilation modes one can control the gas exchange automatically. In terms of CO2-management they use a target minute volume to control end-tidal CO2 and adjust depending on the amount of spontaneously triggered breaths the respiratory rate and the inspiratory pressure support or solely the pressure support. In terms of O2-management according to the peripheral O2 saturation target the PEEP (lung recruitment) and the fraction of inspired oxygen (FiO2) will be set. Both of these controllers depend on an accurate measurement of either end-tidal CO2 and peripheral O2 saturation, respectively.

There exist two recommendations how to ventilate patients with ARDS on an ECMO. First and foremost, the general guidelines of the Extracorporeal Life Support Organization (ELSO) suggest for adults to target a FiO2 of less than 0.3 with a PEEP of 5 to 15 cmH2O and a plateau pressure of less than 25 cm H2O with a respiratory rate of 5 per minute. Whereas Richard et al. in their consensus conference report from 2014 suggest to minimize plateau pressure and PEEP not being specific in terms of numbers. Both guidelines have the goal of keeping the lung at rest concerning patients with ARDS. There are no specific suggestions on ventilation management in patients with heart failure on ECMO. Whether the lung has to be kept open (recruited and less prone to atelectrauma) or kept at rest (less prone to overdistension, either volu- or barotrauma) is at the moment unclear.

Concerning mechanical ventilation settings in patients with ARDS Serpa Neto and colleagues published in 2016 a meta-analysis of nine studies, which included around 550 patients receiving ECMO for refractory hypoxemia. They showed that in these patients driving pressure was associated with in-hospital survival (survivors had a driving pressure of 16.9 cmH2O and non-survivors of 19.4, p 0.004, adjusted HR 1.06 with a 95% CI of 1.03 - 1.10). This is consistent with the study of Amato et al where they showed a reduction of the multivariate relative risk of in-hospital mortality in patients with ARDS - without ECMO - with a driving pressure of less than 15 cmH2O.

The adaptive lung ventilation mode Intellivent-ASV+® has been shown to ventilate normal lungs, lungs with ARDS and COPD within the limits of safe ventilation recommended by the guidelines. Patients on Intellivent-ASV+® had tidal volumes (Vt) ≤ 8 ml/kg/BW, plateau pressure (Pplat) < 30 cmH2O and a driving pressure < 15 cmH2O. Compared to conventional ventilation, patients on Intellivent-ASV+® mode had higher PEEP and lower FiO2, suggesting better recruitment of the dependent part of the lung.

Combining mechanical ventilation using the Intellivent-ASV+® mode and ECMO offers a unique opportunity of having a mechanical ventilator which automatically adapts to lung mechanics and the contribution of ECMO supporting gas exchange.

The main objective of this research project is to propose and verify whether the ventilation mode Intellivent-ASV+® is capable to execute lung protective ventilation despite the presence of an ECMO altering gas exchange.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical Ventilation and ECMO
* Refractory Acute Respiratory Distress Syndrome or Refractory Cardiogenic Shock

Exclusion Criteria:

* Contraindications for ECMO
* Contraindications for Closed Loop Ventilation
* Rejection of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03-06 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

PRIMARY OUTCOMES:
Change in Tidal Volumes | Mixed Model Assessment at baseline (conventional mode), 0 (switch to closed loop), 8, 16, 24, 48 and 72 hours
  Assessment of tidal volumes over the initial 72 hours post switch to closed loop mechanical ventilation
Change in Driving Pressure | Mixed Model Assessment at baseline (conventional mode), 0 (switch to closed loop), 8, 16, 24, 48 and 72 hours
  Assessment of Driving Pressure over the initial 72 hours post switch to closed loop mechanical ventilation
Change in Peak Pressure | Mixed Model Assessment at baseline (conventional mode), 0 (switch to closed loop), 8, 16, 24, 48 and 72 hours
  Assessment of Peak Pressure over the initial 72 hours post switch to closed loop mechanical ventilation
Change in Mechanical Power | Mixed Model Assessment at baseline (conventional mode), 0 (switch to closed loop), 8, 16, 24, 48 and 72 hours
  Assessment of Mechanical Power over the initial 72 hours post switch to closed loop mechanical ventilation
Change in Partial Pressure of Arterial Oxygen | Mixed Model Assessment at baseline (conventional mode), 0 (switch to closed loop), 8, 16, 24, 48 and 72 hours
  Assessment of Partial Pressure of Arterial Oxygen over the initial 72 hours post switch to closed loop mechanical ventilation
Change in Partial Pressure of Arterial CO2 | Mixed Model Assessment at baseline (conventional mode), 0 (switch to closed loop), 8, 16, 24, 48 and 72 hours
  Assessment of Partial Pressure of Arterial CO2 over the initial 72 hours post switch to closed loop mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, Principal Investigator — Medizinische Intensivstation D-HOER 27, UniversitatsSpital Zürich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ELSO Guidelines for Cardiopulmonary Extracorporeal Life Support Extracorporeal Life Support Organization, Version 1.4 August 2017 Ann Arbor, MI, USA
- [Background] Richard C, Argaud L, Blet A, Boulain T, Contentin L, Dechartres A, Dejode JM, Donetti L, Fartoukh M, Fletcher D, Kuteifan K, Lasocki S, Liet JM, Lukaszewicz AC, Mal H, Maury E, Osman D, Outin H, Richard JC, Schneider F, Tamion F. Extracorporeal life support for patients with acute respiratory distress syndrome: report of a Consensus Conference. Ann Intensive Care. 2014 May 24;4:15. doi: 10.1186/2110-5820-4-15. eCollection 2014. PMID 24936342
- [Background] Pesenti A, Carlesso E, Langer T, Mauri T. Ventilation during extracorporeal support : Why and how. Med Klin Intensivmed Notfmed. 2018 Feb;113(Suppl 1):26-30. doi: 10.1007/s00063-017-0384-8. Epub 2017 Nov 28. PMID 29184987
- [Background] Serpa Neto A, Schmidt M, Azevedo LC, Bein T, Brochard L, Beutel G, Combes A, Costa EL, Hodgson C, Lindskov C, Lubnow M, Lueck C, Michaels AJ, Paiva JA, Park M, Pesenti A, Pham T, Quintel M, Marco Ranieri V, Ried M, Roncon-Albuquerque R Jr, Slutsky AS, Takeda S, Terragni PP, Vejen M, Weber-Carstens S, Welte T, Gama de Abreu M, Pelosi P, Schultz MJ; ReVA Research Network and the PROVE Network Investigators. Associations between ventilator settings during extracorporeal membrane oxygenation for refractory hypoxemia and outcome in patients with acute respiratory distress syndrome: a pooled individual patient data analysis : Mechanical ventilation during ECMO. Intensive Care Med. 2016 Nov;42(11):1672-1684. doi: 10.1007/s00134-016-4507-0. Epub 2016 Sep 1. PMID 27586996
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Arnal JM, Wysocki M, Novotni D, Demory D, Lopez R, Donati S, Granier I, Corno G, Durand-Gasselin J. Safety and efficacy of a fully closed-loop control ventilation (IntelliVent-ASV(R)) in sedated ICU patients with acute respiratory failure: a prospective randomized crossover study. Intensive Care Med. 2012 May;38(5):781-7. doi: 10.1007/s00134-012-2548-6. Epub 2012 Mar 30. PMID 22460854
- [Background] Arnal JM, Garnero A, Novonti D, Demory D, Ducros L, Berric A, Donati S, Corno G, Jaber S, Durand-Gasselin J. Feasibility study on full closed-loop control ventilation (IntelliVent-ASV) in ICU patients with acute respiratory failure: a prospective observational comparative study. Crit Care. 2013 Sep 11;17(5):R196. doi: 10.1186/cc12890. PMID 24025234